CLINICAL TRIAL: NCT05449457
Title: Aesthetic Outcome of Layered Closure vs. Layered Closure Followed by 2-Octyl Cyanoacrylate: A Randomized Evaluator-Blinding Split-Wound Comparative Effectiveness Trial
Brief Title: Aesthetic Outcome of Layered Closure vs. Layered Closure Followed by 2-Octyl Cyanoacrylate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 1860725
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2023-06

CONDITIONS: Scarring
MeSH Terms: conditions — Cicatrix | interventions — octyl 2-cyanoacrylate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Two blinded observers will record their scores independently using the POSAS instrument.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Layered Closure (No Intervention): One half of the wound will have a cutaneous layer of sutures (2 layers), as is standard of care, while the other half of the wound will have an additional layer of 2-octyl cyanoacrylate (3 layers).
- Layered Closure with 2-Octyl Cyanoacrylate (Experimental): One half of the wound will have a cutaneous layer of sutures (2 layers), as is standard of care, while the other half of the wound will have an additional layer of 2-octyl cyanoacrylate (3 layers).
  Interventions: Other: 2-Octyl cyanoacrylate

INTERVENTIONS:
Other: 2-Octyl cyanoacrylate — Involves closure supplemented by 2-octyl cyanoacrylate (3 layers)
  Other Names: Dermabond
  Arms: Layered Closure with 2-Octyl Cyanoacrylate

SUMMARY:
Following skin surgeries on the head and neck, several surgeons use a type of surgical glue (such as Dermabond) as a final layer on the top of wound. This glue is thought to seal the wound. Up until this point, there is limited data about the exact advantages or disadvantages of using this glue. We wish to determine if there is a difference in the cosmetic outcome of the scar when the glue is applied compared to when the glue is not applied. In addition, we want to determine if patients prefer to care for a wound with or without the glue.

DETAILED DESCRIPTION:
Sutures are the standard of care in repairing cutaneous wounds. The majority of surgical reconstructions following a Mohs micrographic surgery and standard surgical excisions require two layers of sutures: a deep (subcutaneous) layer and a superficial (cuticular) layer.

Alternatively, skin adhesives, such as 2-octyl cyanoacrylate (commercially available as "Dermabond"), have been used successfully in lieu of the outer layer of sutures. Cosmetic outcomes with 2-octyl cyanoacrylate have been shown to be equivalent to sutured wounds, perhaps with a lower infection rate. However, wounds repaired with 2-octyl cyanoacrylate may have a higher dehiscence rate.

Recently, surgeons have been using 2-octyl cyanoacrylate, in addition to dissolvable sutures. This is thought to combine the advantages of 2-octyl cyanoacrylate, including easier wound care and lower infection rate, with the lower dehiscence rate of sutures.

A previous study by Zhuang et al found no difference in wound cosmesis between deep sutures supplemented by 2-octyl cyanoacrylate compared with layered closure with 5-0 fast-absorbing gut suture, with the exception of inferior scar pigmentation with 2-octyl cyanoacrylate.1 Several studies likewise found no significant differences between 2-octyl cyanoacrylate versus sutures in repairing cutaneous wounds.

To our knowledge, no study has been conducted directly comparing closure (2 layers) versus closure supplemented by 2-octyl cyanoacrylate (3 layers). We hope that our study will provide new insight into this aspect of cutaneous surgery.

ELIGIBILITY:
All patients scheduled for cutaneous surgical procedures with one of the study investigators at the UC Davis Dermatology Clinic will be screened for eligibility.

Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure on the face or neck with predicted primary closure.
* Willing to return for follow up visit

Exclusion Criteria:

* Incarceration
* Under 18 years of age
* Pregnant women
* Unable to understand written and oral English.
* Wounds with predicted closure length less than 3 cm

None of these special populations will be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Scar Assessment as measured by Patient Observer Scar Assessment Score (POSAS) | 3 months
  The primary endpoint will be the score of two blinded reviewers independently using the POSAS assessment. The observer scale of the POSAS consists of six items (vascularity, pigmentation, thickness, relief, pliability, and surface area). All items are scored on a scale ranging from 1 ("like normal skin") to 10 ("worst scar imaginable"). The sum of the six items results in a total score of the POSAS observer scale. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10. All parameters should preferably be compared to normal skin on a comparable anatomic location.
Width of Scar as measured using Trace-to-Tape Method | 3 months
  The trace-to-tape method is an objective measure for linear postoperative scars. The mean scar width will be determined using the trace-to-tape method. The surface area of the scar will be collected by tracing the scar with a water-based gel pen. While still wet, the gel residue will be lifted from the skin with clear packing tape and transferred on a sheet of paper.

SECONDARY OUTCOMES:
Complications or Adverse Events from Treatment | 3 months
  For example, if one half of the scar has more associated erythema, as measured using the Trace-to-Tape method, then it will be recorded. Other complications from the treatment will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis - Dermatology Department, Sacramento, California, United States